CLINICAL TRIAL: NCT06537856
Title: The Effect of Health Education Based on Health Belief Model and Text Messages Given to Firefighters on The Level of Knowledge, Awareness and Quality Of Life About Cardiovascular Disease Risk Factors
Brief Title: Impact of Education and Text Messages on Cardiovascular Disease Risk Factors Awareness Knowledge and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Zehra Kartoğlu, Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MU-HSI-ZK-01
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases
Keywords: Health Belief Model; Firefighter; Occupational Health Nursing; Cardiovascular disease; Risk Factors; Health Education
MeSH Terms: conditions — Cardiovascular Diseases; Health Education

STUDY DESIGN:
Intervention Model Description: In the study, there are two parallel groups as control and intervention groups
Who Masked: Participant
Masking Description: In the study, participant blinding was performed by ensuring that the participants did not know which group they were in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Prior to the intervention, both the control and intervention groups were interviewed face-to-face and completed the Cardiovascular Disease Risk Awareness Rating Scale (CDRAAS), the Cardiovascular Disease Risk Factor Knowledge Level Scale (CARRF-KL) and the EQ-5D Quality of Life Scale. The intervention group then received health belief model-based cardiovascular disease risk factor prevention training. This training, conducted by the researcher, was carried out in 3 sessions, including interactive question-answer sessions. After the training, a total of 39 reminder text messages were sent to the intervention group via WhatsApp 2-3 times a week for 12 weeks.
  Interventions: Other: Health Belief Model Based Cardiovascular Disease Risk Factor Prevention Education; Behavioral: Reminder Short Messages
- No intervention (No Intervention): No intervention was given to the control group. After the education given to the intervention group and the reminder text messages sent for 12 weeks, the intervention and control groups were asked to fill out the Cardiovascular Disease Risk Awareness Rating Scale (CDRAAS), Cardiovascular Disease Risk Factor Knowledge Level Scale (CARRF-KL) and EQ-5D Quality of Life Scale again in the same week. After the post-tests were taken, the control group also received training.

INTERVENTIONS:
Other: Health Belief Model Based Cardiovascular Disease Risk Factor Prevention Education — In line with the literature review, "Health Belief Model-Based Cardiovascular Disease Risk Factor Prevention Training" was created in order to increase the level of knowledge of firefighters regarding cardiovascular disease risk factors, improve their awareness and positively affect their quality of life. This training was given in 3 different sessions by meeting face-to-face with firefighters in the training hall of the fire stations. Each session lasted 40 minutes. Answers were given to the questions asked at the end of the session. The training was organized under the following main headings:
  Perceived Sensitivity, Perceived Seriousness, Perceived Barriers, Perceived Self-Efficacy, Health Motivation/Activators
  Other Names: Reminder Short Messages
  Arms: Intervention
Behavioral: Reminder Short Messages — After the Health Belief Model-Based health education, 39 text messages were sent via WhatsApp application 3-4 times a week for 3 months to increase the effectiveness of the education and the motivation of firefighters in CVD prevention.
  Arms: Intervention

SUMMARY:
This study was planned to evaluate the effect of a health education program based on the health belief model and text messages on the level of knowledge, awareness and quality of life regarding cardiovascular disease risk factors in firefighters. A total of 160 firefighters, 84 in the intervention group and 76 in the control group, constituted the sample of the study.

Hypotheses of the Study H1 The mean CDRAAS posttest scores of the firefighters in the intervention group after health education will be higher than the mean posttest scores of the control group.

H2 The mean CDRAAS post-test scores of the firefighters in the intervention group after the health education will be higher than the mean pre-test scores.

H3 The mean CARRIF-KL posttest scores of the firefighters in the intervention group after health education will be higher than the mean posttest scores of the control group.

H4 The mean CARRIF-KL posttest scores of the firefighters in the intervention group after the health education will be higher than the mean pretest scores.

H5 The mean EQ-5D posttest scores of the firefighters in the intervention group after health education will be higher than the mean posttest scores of the control group.

H6 The mean EQ-5D posttest scores of the firefighters in the intervention group after health education will be higher than the mean pretest scores.

DETAILED DESCRIPTION:
In this study, a randomized control group pretest-posttest design was used to evaluate the effect of a health education program based on the health belief model and text messages on the level of knowledge, awareness and quality of life regarding cardiovascular disease risk factors in firefighters.

The power analysis was applied based on a 5% significance level (or 95% confidence interval), two-way, 80% power requirement. As a result of the analysis, the minimum sample size required for each group (intervention and control) in the study was calculated as 67 people. The intervention group received health education on prevention of cardiovascular disease risk factors based on the Health Belief Model consisting of 3 sessions. Following the health education, a total of 39 reminder text messages were sent via WhatsApp three or four times a week for 12 weeks to increase self-efficacy and health motivation. Data were collected through face-to-face interviews and by using the Cardiovascular Disease Risk Awareness Rating Scale, the Cardiovascular Disease Risk Factor Knowledge Level Scale and the EQ-5D Quality of Life Scale. In data analysis, dependent samples t test (paired samples t test) was used for intra-group mean comparisons and independent samples t test (independent samples t test) was used for inter-group mean comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* No reading and comprehension problems,
* Individuals who agreed to participate in the study,
* Not having any cardiovascular disease,
* To be working in the institution where the research is carried out,
* Not having any mental illness or a disease/disabily that would prevent working ,
* Not having any structured training in preventing cardiovascular disease.

Exclusion Criteria:

* Under 18,
* Having cardiovascular disease,
* Refuses to work or wants to leave during the work,
* Individuals with reading and comprehension problems,
* To have received any training on cardiovascular disease prevention,
* Having any mental illness or disease/disability that would prevent participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Disease Risk Awareness Assessment Scale (CDRAAS) | two weeks
  The scale consists of three sub-dimensions: perceived heart attack/stroke risk, perceived benefits and intentions to change, and healthy eating intentions. The scale, which consists of 22 items in total, is a 4-point Likert scale and is scored between 1 (strongly disagree) and 4 (strongly agree). Higher scale and subscale scores indicate increased awareness of cardiovascular diseases.

SECONDARY OUTCOMES:
The Cardiovascular Disease Risk Factors Knowledge Level (CARRF-KL) | two weeks
  The scale is used to measure the level of knowledge about cardiovascular disease risk factors. While the first four items in the scale are related to the characteristics of cardiovascular diseases, preventability and age factor, 15 items question risk factors and nine items question the result of change in risk behaviors. Scale items are answered with 'True', 'False' and 'Don't know' options. Each correct answer is scored as 1 point. Scores that can be obtained from the scale vary between 0 and 28, with the highest score being 28 and the lowest score being 0. The higher the score obtained from the scale, the higher the level of knowledge.
EuroQol Quality of Life Scale | two weeks
  It is a quality of life scale that measures how individuals perceive and evaluate their own health status. The scale consists of two parts: EQ-5D Index and EQ-5D (Visual Analog Score (VAS). EQ-5D index: It consists of 5 dimensions: movement, pain, general activities, self-care, anxiety/depression. The answers to each dimension have 5 options: no problem, mild problem, moderate problem, severe problem and extreme problem. EQ-5D VAS: It is a visual analog scale in which individuals give values between 0 and 100 about their current health status and mark it on a thermometer-like scale. Quality of life scores ranging from 0 to 100 are obtained with the scale. An increase in the scale score indicates a positive perception of health.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kartoğlu, M.Sc Student, Principal Investigator — zehra.kartoglu@aljazari.k12.tr
Locations (1):
- Aljazari International School of Science and Technology, Istanbul, Atakent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No